CLINICAL TRIAL: NCT06205212
Title: The Effect of High-flow Nasal Cannula Applied During Preoxygenation for Prevention of Atelectasis in Patients With Obesity Undergoing General Anesthesia: A Randomized Controlled Trial
Brief Title: High-flow Nasal Oxygenation During Preoxygenation and Atelectasis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: SMG-SNU Boramae Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: HFNO_PRE
Record Dates: First submitted 2023-09-19; First posted 2024-01-12 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2023-09

CONDITIONS: Anesthesia, General; Pulmonary Atelectasis
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- facemask (Active Comparator): preoxygenation using a conventional facemask
  Interventions: Other: facemask
- high-flow nasal oxygen (Experimental): preoxygenation using high-flow nasal cannula oxygen
  Interventions: Other: high-flow nasal oxygen

INTERVENTIONS:
Other: high-flow nasal oxygen — preoxygenation using high-flow nasal oxygen, FiO2 1.0, 40 L/min, 3 min
  Arms: high-flow nasal oxygen
Other: facemask — preoxygenation using facemask, FIO2 1.0, fresh gas flow 10 L/min, 3 min
  Arms: facemask

SUMMARY:
Atelectasis after induction of general anesthesia is common even in healthy patients and is clinically problematic, especially in obese patients. We aim to investigate whether preoxygenation with high-flow nasal oxygen during anesthesia induction reduces atelectasis in obese patients.

ELIGIBILITY:
Inclusion Criteria:

* Adults patients undergoinig surgery under general anesthesia with a BMI of 30 kg/m2 or greater who have given informed consent

Exclusion Criteria:

* surgery time less than 2 hours
* Nasotracheal intubation
* Severe cardiac or respiratory disease
* History of difficult airway
* History of a surgery or anatomical anomaly in the head and neck
* History of Inability to breathe through nose
* Gastric reflux disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2023-10-10 (Actual); Primary Completion 2024-10-10 (Estimated); Study Completion 2024-10-10 (Estimated)

PRIMARY OUTCOMES:
Lung ultrasound score | Immediately after anesthesia induction
  modified LUSS

SECONDARY OUTCOMES:
Incidence of atelectasis | Immediately after anesthesia induction
PaO2 to FiO2 ratio and PaCO2 | Immediately after anesthesia induction
Hemodynamic variables | During anesthesia induction
  Blood pressure, heart rate, pulse oximetry
Patient Satisfaction Score | During preoxygenation
Lung ultrasound score | In the PACU after surgery
Incidence of Spo2 less than 95% | during 48 hours postoperatively
Maximum body temperature | during hospitalization up to 1 week
Incidence of postoperative pulmonary complications | during hospitalization up to 1 week
length of hospital stay | up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: TAE KYONG KIM, Principal Investigator — SMG-SNU Boramae Medical Center
Locations (1):
- SMG - SNU Boramae Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No